CLINICAL TRIAL: NCT02618902
Title: A "negative"dendritic Cell-based Vaccine for the Treatment of Multiple Sclerosis: a First-in-human Clinical Trial
Acronym: MS-tolDC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Zwi Berneman, Professor, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCRG15-001
Record Dates: First submitted 2015-11-18; First posted 2015-12-02 (Estimated); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis
Keywords: patient safety; tolerogenic dendritic cells; tolDC
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- tolerogenic dendritic cells (tolDC) (Experimental): Each vaccine (5x106, 10x106 , or 15x106cells in 500 µL NaCl 0.9% solution supplemented with 5% human albumin) will be administered through intradermal injection at 5 sites (100 µL/site) in the subclavicular region (5-10 cm from the cervical lymph nodes). Injection sites will alternate between left and right sides.
  Interventions: Biological: tolerogenic dendritic cells (tolDC)

INTERVENTIONS:
Biological: tolerogenic dendritic cells (tolDC) — dose-escalation

SUMMARY:
A first-in-human clinical trial to treat patients with multiple sclerosis by vaccination with tolerogenic dendritic cells (tolDC), generated using Good Manufacturing Practice (GMP) will be conducted. In doing so, the feasibility and safety of administering myelin-derived peptide-pulsed tolDC in patients with MS will be assessed.

DETAILED DESCRIPTION:
A phase I dose-escalating clinical trial will be conducted in a coordinated and comprehensive manner to determine safety and tolerability, and to enable selection of a suitable dose regimen for phase II trials. The primary objective of the phase I study will be to determine whether tolDC-based therapy is safe and well tolerated and to establish the dose-response, with clinical relapse rates, neurological disability (assessed using various scales) and MRI endpoints, measured over 12 months. Patients will serve as their own controls pre- and post-vaccination. Completion of screening assessments and confirmation of eligibility criteria should take no longer than 6 weeks. First-line treatments will be stopped 6 weeks before baseline at the latest.

ELIGIBILITY:
Inclusion Criteria:

* MS according to 2010 revised McDonald criteria (76);
* Expanded disability status scale (EDSS) of 0-6.5 inclusive;
* Disease duration of maximum 15 years and first signs or symptoms at least 6 months prior to enrolment in the study;
* Active MS (relapsing and progressive): -1 relapse in the past year and/or

  * at least 1 enhancing lesion on brain MRI in the past year
  * new or enlarging T2 lesion(s) in comparison with a reference scan from maximum 1 year before
* Neurologically stable with no evidence of relapse for at least 30 days prior to start of screening and throughout during the screening phase;
* Positive T cell reactivity response to a mix of 7 myelin-derived peptides;
* Able to sign informed consent;
* Ability to comply with the protocol assessments;
* Appropriate venous access.
* Use of adequate contraceptive measures

Exclusion Criteria:

* Previous use of immunosuppressive or cytostatic treatment, including mitoxantrone, alemtuzumab or bone marrow transplantation or stem cell transplantation at any time prior to enrolment;
* Treatment with fingolimod or natalizumab or dimethylfumarate or teriflunomide within the last 3 months prior to study enrolment;
* Pregnancy or planning pregnancy in the next 12 months and breast feeding;
* Drug or alcohol abuse;
* Inability to undergo MRI assessments;
* History of or actual signs of immunodeficiency or malignancies;
* Concurrent clinically relevant cardiac, immunological, pulmonary, neurological, renal or other major disease;
* Hepatitis B, C, HIV, Syphilis or tuberculosis
* Splenectomy;
* Dementia or severe psychiatric, cognitive or behavioral problems or other comorbidity that could interfere with the compliance to the protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Safety (Occurrence and severity of adverse events will be recorded) | 6 months
  Occurrence and severity of adverse events will be recorded
Feasibility (Generation of GMP-grade cell product released according to QC) | 6 months
  Generation of GMP-grade cell product released according to QC

SECONDARY OUTCOMES:
Expanded disability status scale (EDSS) | 6 months
  The patients' disability level well be checked during every visit
9 Hole Peg Test (9HPT) | 6 months
  This is a brief, standardized, quantitative test of upper extremity function
25 Foot walk test (T25FW) | 6 months
  This is a quantitative mobility and leg function performance test based on a timed 25-walk.
Symbol Digit Modalities test (SDMT) | 6 months
  This test quickly screens for organic cerebral dysfunction
Number of Gd-enhancing lesions on MRI | 6 months
  By means of MRI Gd-enhancing lesions will be analysed
Number of new or enlarging T2 lesions on MRI | 6 months
  By means of MRI new or enlarging T2 lesions will be analysed

OTHER OUTCOMES:
MSQOL-54 | 6 months
  The MSQOL-54 is a multidimensional health-related quality of life measure that combines both generic and MS-specific items into a single instrument
whole-blood lymphocyte phenotyping - immunomonitoring | 6 months
  Blood samples will be analysed into detail, before and after completion of the vaccination cycle
cytokine profiling - immunomonitoring | 6 months
  Blood samples will be analysed into detail, before and after completion of the vaccination cycle
pathogenic T cell responses - immunomonitoring | 6 months
  myelin-specific T cell reactivity will be determined before and after completion of the vaccination cycle

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Cools, PhD, Principal Investigator — Universiteit Antwerpen; Zwi Berneman, MD, PhD, Study Director — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Belgium

REFERENCES:
- [Derived] Willekens B, Presas-Rodriguez S, Mansilla MJ, Derdelinckx J, Lee WP, Nijs G, De Laere M, Wens I, Cras P, Parizel P, Van Hecke W, Ribbens A, Billiet T, Adams G, Couttenye MM, Navarro-Barriuso J, Teniente-Serra A, Quirant-Sanchez B, Lopez-Diaz de Cerio A, Inoges S, Prosper F, Kip A, Verheij H, Gross CC, Wiendl H, Van Ham MS, Ten Brinke A, Barriocanal AM, Massuet-Vilamajo A, Hens N, Berneman Z, Martinez-Caceres E, Cools N, Ramo-Tello C; RESTORE consortium. Tolerogenic dendritic cell-based treatment for multiple sclerosis (MS): a harmonised study protocol for two phase I clinical trials comparing intradermal and intranodal cell administration. BMJ Open. 2019 Sep 9;9(9):e030309. doi: 10.1136/bmjopen-2019-030309. PMID 31501122